CLINICAL TRIAL: NCT06855927
Title: The Effect of Guided Imagery on Activity-Specific Balance Confidence, Pain, and Psychological Well-Being in Elderly Orthopedic Patients: A Randomized Controlled Trial
Brief Title: The Effect of Guided Imagery on Activity-Specific Balance Confidence, Pain, and Psychological Well-Being
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Neslihan Söylemez, PhD, Research Assistant, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: Osmaniye Korkut Ata University
Record Dates: First submitted 2025-02-25; First posted 2025-03-04 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Guided Imagery
Keywords: Orthopedics; Guided Imagery; pain; Psychological Well-Being
MeSH Terms: conditions — Pain; Psychological Well-Being | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Effect of Guided Imagery in Elderly Orthopedic Patients (Experimental): Guided imagery, which is a mind-body method, allows the patient to relax and feel good. In this way, patients' self-confidence increases.
  Interventions: Other: Guided Imagery
- Balance Confidence, Pain, and Psychological Well-Being in Elderly Orthopedic Patients (No Intervention): No intervention is applied to the patients in this group and the effectiveness of the interventions used on the patients in the other group is measured.

INTERVENTIONS:
Other: Guided Imagery — Guided imagery is a potential healing technique that aims to help individuals mentally visualize positive physical and psychological states.
  Other Names: Dreaming
  Arms: The Effect of Guided Imagery in Elderly Orthopedic Patients

SUMMARY:
The aim of this clinical trial is to evaluate the effect of guided imagery on activity-specific balance confidence, pain, and psychological well-being in elderly orthopedic patients. In the study, guided imagery will be applied by the researchers and will be applied over 2 days for a total of 3 repetitions. The study will be conducted in the postoperative period of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are open to communication and collaboration,
* Those who are over 65 years old,
* Those who have a mini-mental test score of 24 and above,
* Those who have the same type of analgesic protocol,
* Those who have a numerical pain score of at least 4 will be included.

Exclusion Criteria:

* Patients who have developed any complications,
* Patients who have hearing, vision and perception problems,
* Patients who have been diagnosed with any psychiatric disease,
* Patients who have developed any complications after surgery will be excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Guided imagery applied to elderly orthopedic patients increases activity-specific balance confidence. | 100 minutes
  The patient relaxes as a result of guided imagery, activity-specific balance confidence will be measured with the Activity-Specific Balance Confidence Scale. The scale is based on ratings of perceived balance level during different activities of daily living from 0% (no confidence) to 100% (full confidence). The total score ranges from 0 to 100. Higher scores indicate greater confidence. The intervention will be evaluated 3 times. 39 patients will be measured in the touch group.
Guided imagery applied to elderly orthopedic patients reduces pain levels. | 100 minutes
  The patient is relaxed as a result of guided imagery, the pain value will be measured with a verbal pain scale. On this scale, 0 describes the absence of pain, while 10 describes the highest level of pain, which is unbearable. Higher scores indicate more pain. The intervention will be evaluated 3 times. 39 patients will be measured in the touch group.
Guided imagery applied to elderly orthopedic patients increases psychological well-being. | 100 minutes
  The patient relaxes as a result of guided imagery, and the level of psychological well-being will be measured with the Psychological Well-being Scale. The total scale score varies between 8 and 56. As the total scale score increases, the level of psychological well-being also increases. The intervention will be evaluated 3 times. 39 patients will be measured in the touch group.

CONTACTS AND LOCATIONS:
Overall Officials: Adile Bozkurt Tonguç, PhD, Study Chair — Osmaniye Korkut Ata University